CLINICAL TRIAL: NCT03452397
Title: Multicenter, Randomized, Controlled, Double-Masked Clinical Trial to Evaluate the Efficacy of OC-02 Nasal Spray on Signs and Symptoms of Dry Eye Disease (The PEARL Study)
Brief Title: Clinical Trial to Evaluate the Efficacy of OC-02 Nasal Spray on Signs and Symptoms of Dry Eye Disease (The PEARL Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPP-001
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 0.2 % hemigalactarate (0.11% free base) 0.2 % OC-02 Low Dose (1.1 mg/mL) (Active Comparator): 0.2 % hemigalactarate (0.11% free base) 0.2 % OC-02 Low Dose (1.1 mg/mL)
  Interventions: Drug: 0.2 % hemigalactarate (0.11% free base) 0.2 % OC-02 Low Dose (1.1 mg/mL)
- 1.0 % hemigalactarate (0.11% free base) 1.0 % OC-02 Mid Dose (5.5 mg/mL) (Active Comparator): 1.0 % hemigalactarate (0.11% free base) 1.0 % OC-02 Mid Dose (5.5 mg/mL)
  Interventions: Drug: 1.0 % hemigalactarate (0.11% free base) 1.0 % OC-02 Mid Dose (5.5 mg/mL)
- 2.0 % hemigalactarate (0.11% free base) 2.0 % OC-02 High Dose (11.1 mg/mL) (Active Comparator): 2.0 % hemigalactarate (0.11% free base) 2.0 % OC-02 High Dose (11.1 mg/mL)
  Interventions: Drug: 2.0 % hemigalactarate (0.11% free base) 2.0 % OC-02 High Dose (11.1 mg/mL)
- Placebo (vehicle) nasal spray (Placebo Comparator): Placebo (vehicle) nasal spray
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: 0.2 % hemigalactarate (0.11% free base) 0.2 % OC-02 Low Dose (1.1 mg/mL) — 0.2 % hemigalactarate (0.11% free base) 0.2 % OC-02 Low Dose (1.1 mg/mL)
  Arms: 0.2 % hemigalactarate (0.11% free base) 0.2 % OC-02 Low Dose (1.1 mg/mL)
Drug: 1.0 % hemigalactarate (0.11% free base) 1.0 % OC-02 Mid Dose (5.5 mg/mL) — 1.0 % hemigalactarate (0.11% free base) 1.0 % OC-02 Mid Dose (5.5 mg/mL)
  Arms: 1.0 % hemigalactarate (0.11% free base) 1.0 % OC-02 Mid Dose (5.5 mg/mL)
Drug: 2.0 % hemigalactarate (0.11% free base) 2.0 % OC-02 High Dose (11.1 mg/mL) — 2.0 % hemigalactarate (0.11% free base) 2.0 % OC-02 High Dose (11.1 mg/mL)
  Arms: 2.0 % hemigalactarate (0.11% free base) 2.0 % OC-02 High Dose (11.1 mg/mL)
Drug: Placebo (vehicle) nasal spray — Placebo (vehicle) nasal spray
  Arms: Placebo (vehicle) nasal spray

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of OC-02 Nasal Spray as compared to placebo on signs and symptoms of dry eye disease.

DETAILED DESCRIPTION:
This was a Phase 2, multicenter, randomized, double-masked, placebo controlled study designed to evaluate the safety and efficacy of OC 02 Nasal Spray in adult participants with dry eye disease. Approximately 160 subjects, at least 22 years of age, with a subject-reported history of dry eye disease and meeting all other study eligibility criteria were planned to be randomized to receive an application of OC-02 or placebo at Visit 1 and Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to Visit 1

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery), extraocular surgery (such as blepharoplasty) in either eye within three months or refractive surgery within twelve months of Visit 1
* Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with DED are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Louisville, Louisville, Kentucky
  - Andover, Andover, Massachusetts
  - Nashville, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torkildsen GL, Pattar GR, Jerkins G, Striffler K, Nau J. Efficacy and Safety of Single-dose OC-02 (Simpinicline Solution) Nasal Spray on Signs and Symptoms of Dry Eye Disease: The PEARL Phase II Randomized Trial. Clin Ther. 2022 Sep;44(9):1178-1186. doi: 10.1016/j.clinthera.2022.07.006. Epub 2022 Aug 11. PMID 35965109

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.2% Hemigalactarate (0.11% Free Base) 0.2% OC-02 Mid Dose (1.1 mg/mL): 0.2% hemigalactarate (0.11% free base) 0.2% OC-02 Mid Dose (1.1 mg/mL)
- 1% Hemigalactarate (0.11% Free Base) 1% OC-02 Mid Dose (5.5 mg/mL): 1% hemigalactarate (0.11% free base)
  1% OC-02 Mid Dose (5.5 mg/mL)
- 2% Hemigalactarate (0.11% Free Base) 2% OC-02 High Dose (11.1 mg/mL): 2% hemigalactarate (0.11% free base) 2% OC-02 High Dose (11.1 mg/mL)
Period: Overall Study
Arm/Group | 0.2% Hemigalactarate (0.11% Free Base) 0.2% OC-02 Mid Dose (1.1 mg/mL) | 1% Hemigalactarate (0.11% Free Base) 1% OC-02 Mid Dose (5.5 mg/mL) | 2% Hemigalactarate (0.11% Free Base) 2% OC-02 High Dose (11.1 mg/mL) | Placebo (Vehicle) Nasal Spray
Started | 41 | 41 | 41 | 42
Completed | 40 | 41 | 39 | 41
Not Completed | 1 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Administrative reason | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects in the ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.2 % Hemigalactarate (0.11% Free Base) 0.2 % OC-02 Low Dose (1.1 mg/mL) | 1.0 % Hemigalactarate (0.11% Free Base) 1.0 % OC-02 Mid Dose (5.5 mg/mL) | 2.0 % Hemigalactarate (0.11% Free Base) 2.0 % OC-02 High Dose (11.1 mg/mL) | Placebo (Vehicle) Nasal Spray | Total
Number analyzed (Participants) | 41 | 41 | 41 | 42 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (11.80) | 64.0 (11.15) | 62.7 (9.30) | 64.4 (11.76) | 63.9 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 31 | 34 | 118
  Male | 17 | 12 | 10 | 8 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic/Latino | 41 | 40 | 41 | 39 | 161
  Not reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Alaskan Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 0 | 3
  Black/African American | 3 | 2 | 3 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 37 | 37 | 37 | 39 | 150
  Multiple races | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 41 | 42 | 165

OUTCOME MEASURES:

1. Primary Outcome: Schirmer's Test Score at Day 1
Description: The primary endpoint was the change in anesthetized Schirmer's Test Score (STS) from baseline to Day 1. Change in Schirmer test score pre to post treatment. The Schirmer's test measures the amount of tears produced by placing a paper strip in the eye for 5 minutes and distance of wetting was recorded. Schirmer's test scores from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: Day 1 (Pre to Post-Treatment Change)
Population: Subjects in the ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | 0.2 % Hemigalactarate (0.11% Free Base) 0.2 % OC-02 Low Dose (1.1 mg/mL) | 1.0 % Hemigalactarate (0.11% Free Base) 1.0 % OC-02 Mid Dose (5.5 mg/mL) | 2.0 % Hemigalactarate (0.11% Free Base) 2.0 % OC-02 High Dose (11.1 mg/mL) | Placebo (Vehicle) Nasal Spray
Number analyzed (Participants) | 41 | 41 | 41 | 42
mm | 9.0 [6.3 to 11.6] | 17.5 [14.8 to 20.2] | 19.6 [16.9 to 22.3] | 3.0 [0.3 to 5.6]

2. Primary Outcome: Eye Dryness Score at Visit 2
Description: Change in Eye Dryness score from baseline to Day 15. Eye dryness score on a Visual Analogue Scale (VAS) from 0 (no discomfort) to 100 (maximum discomfort) millimeters where a lower score is indicative of a better outcome.
Time Frame: Day 15 (Pre to Post-Treatment Change)
Population: Subjects in the ITT Population. Only Subjects who had both pre-treatment and post-treatment values were utilized in the change from pre-treatment statistics
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Groups:
- 1 % Hemigalactarate (0.11% Free Base) 1 % OC-02 Mid Dose (5.5 mg/mL): 1 % hemigalactarate (0.11% free base)
  1 % OC-02 Mid Dose (5.5 mg/mL)
- 2 % Hemigalactarate (0.11% Free Base) 2 % OC-02 High Dose (11.1 mg/mL): 2 % hemigalactarate (0.11% free base) 2 % OC-02 High Dose (11.1 mg/mL)
Arm/Group | 0.2 % Hemigalactarate (0.11% Free Base) 0.2 % OC-02 Low Dose (1.1 mg/mL) | 1 % Hemigalactarate (0.11% Free Base) 1 % OC-02 Mid Dose (5.5 mg/mL) | 2 % Hemigalactarate (0.11% Free Base) 2 % OC-02 High Dose (11.1 mg/mL) | Placebo (Vehicle) Nasal Spray
Number analyzed (Participants) | 37 | 41 | 38 | 41
mm | -9.4 [-15.4 to -3.5] | -17.4 [-23.1 to -11.7] | -20.7 [-26.7 to -14.7] | -6.5 [-12.1 to -0.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study drug administration until the final study visit at Visit 2, up to 15 days.
Arm/Group | 0.2 % Hemigalactarate (0.11% Free Base) 0.2 % OC-02 Low Dose (1.1 mg/mL) | 1.0 % Hemigalactarate (0.11% Free Base) 1.0 % OC-02 Mid Dose (5.5 mg/mL) | 2.0 % Hemigalactarate (0.11% Free Base) 2.0 % OC-02 High Dose (11.1 mg/mL) | Placebo (Vehicle) Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/41 | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 17/41 | 23/41 | 24/41 | 4/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.2 % Hemigalactarate (0.11% Free Base) 0.2 % OC-02 Low Dose (1.1 mg/mL) (N=41) | 1.0 % Hemigalactarate (0.11% Free Base) 1.0 % OC-02 Mid Dose (5.5 mg/mL) (N=41) | 2.0 % Hemigalactarate (0.11% Free Base) 2.0 % OC-02 High Dose (11.1 mg/mL) (N=41) | Placebo (Vehicle) Nasal Spray (N=42)
failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.2 % Hemigalactarate (0.11% Free Base) 0.2 % OC-02 Low Dose (1.1 mg/mL) (N=41) | 1.0 % Hemigalactarate (0.11% Free Base) 1.0 % OC-02 Mid Dose (5.5 mg/mL) (N=41) | 2.0 % Hemigalactarate (0.11% Free Base) 2.0 % OC-02 High Dose (11.1 mg/mL) (N=41) | Placebo (Vehicle) Nasal Spray (N=42)
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Keratits (Eye disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 15 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 10 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Instillation site irritation (General disorders) | 3 | 4 | 6 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Gastrooesphageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03452397/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03452397/SAP_001.pdf